CLINICAL TRIAL: NCT02424565
Title: An Exploratory Study to Assess the Effect of Topical Application of Iodex® Balm on Local Surface Temperature Using Infra Red Thermal Imaging Technique
Brief Title: Effect of Topical Application of Iodex® Balm on Local Surface Temperature
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 204663
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): 2 ± 0.2 g of product will be gently rubbed for 15 seconds on the affected knee joint.
  Interventions: Drug: IODEX® balm
- Placebo (Placebo Comparator): 2 ± 0.2 g of product will be gently rubbed for 15 seconds on the affected knee joint.
  Interventions: Other: Placebo balm

INTERVENTIONS:
Drug: IODEX® balm — 2 ± 0.2 g of test balm will be applied topically in a crossover fashion at a gap of 3 days between the two product applications.
  Arms: Test
Other: Placebo balm — 2 ± 0.2 g of placebo balm will be applied topically in a crossover fashion at a gap of 3 days between the two product applications.
  Arms: Placebo

SUMMARY:
The rationale of this study is to map out changes in temperature distribution brought about by topical application of our test product, and use this physiological phenomenon to visualize the onset of action involved in overall mechanism of action of the product.

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from chronic osteoarthritis of knee joint (as per American College of Rheumatology criteria) for > 3 months
* Participants in good general and mental health with no clinically significant and relevant abnormalities of medical history or physical examination

Exclusion Criteria:

* Women of child bearing potential, pregnant and lactating women
* Intolerance/hypersensitivity to study material/ingredient
* Recent history of alcohol or drug abuse
* Participants receiving topical non-steroidal antiinflammatory drugs (NSAIDs), other topical analgesics/counterirritants/mineral oils, or other medication, which might interfere with study results
* Participants having psoriasis/active atopic dermatitis/eczema/skin infected lesions/burn/wound at the site of application

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Indiranagar, Banglador, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in India.
Pre-assignment Details: Of the 19 participants screened, 15 were randomized, 14 completed the study.
Groups:
- First Test Balm Then Placebo Balm: 2 ± 0.2 g of test balm of 9g balm packed in each primary package was gently rubbed for 15 seconds on the affected knee joint, then a gap of 3 days as a washout period, followed by application of 2 ± 0.2 g of placebo balm of 9g balm packed in each primary package .
- First Placebo Balm Then Test Balm: 2 ± 0.2 g of placebo balm of 9g balm packed in each primary package was gently rubbed for 15 seconds on the affected knee joint, then a gap of 3 days as a washout period, followed by application of 2 ± 0.2 g of test balm of 9g balm packed in each primary package .
Period: Period 1 (D0)
Arm/Group | First Test Balm Then Placebo Balm | First Placebo Balm Then Test Balm
Started | 8 | 7
Completed | 8 | 6
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Washout Period
Arm/Group | First Test Balm Then Placebo Balm | First Placebo Balm Then Test Balm
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0
Period: Period 2 (D3)
Arm/Group | First Test Balm Then Placebo Balm | First Placebo Balm Then Test Balm
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures is presenting the data of Intent to treat (ITT) population.
Groups:
- Overall Participants: Total number of participants randomized and treated in the study.
Arm/Group | Overall Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Significant Increase in Local Surface Temperature
Description: Local surface temperature was measured by the spectral order of colour after application of product. Infra-red camera was used to take 11 images with one just before application of product and remaining 10 images at every minute for first 10 minutes after application of product. IR camera converted the IR energy radiated by the body into electrical impulses, which were then digitally indicated on a spatial temperature map. IR camera represents the temperature distribution in a so-called rainbow or spectral order of colors. The predominant colour will be determined on a 5 point scale based on Thermal Images produced using Infra-Red Thermography (IRT) technique and recorded as either Blue, Green, Yellow, Orange or Deep Orange/Red (In increasing order of temperature). There was an approximate temperature difference of 0.5°C between adjacent colours on the map which was supposed to brought about by application of the product and considered significant.
Time Frame: Every minute from baseline to 10 minutes
Population: Intent-to-treat (ITT) population included all participants of safety population with any post-treatment assessment. Since no significant increase in surface temperature was observed in subjects for either treatment, therefore, number of subjects analyzed for this outcome is zero.
Groups:
- Test Balm: 2 ± 0.2 g of test balm of 9 g balm packed in each primary package was gently rubbed for 15 seconds on the affected knee joint.
- Placebo Balm: 2 ± 0.2 g of placebo balm of 9 g balm packed in each primary package was gently rubbed for 15 seconds on the affected knee joint.
Arm/Group | Test Balm | Placebo Balm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From application of investigational product upto 5 days.
Groups:
- Placebo Balm: 2 ± 0.2 g of placebo balm of 9g balm packed in each primary package was gently rubbed for 15 seconds on the affected knee joint.
Arm/Group | Test Balm | Placebo Balm
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
Primary outcome measure was to detect significant increase in surface temperature. Since this was not observed for either treatment, there was no statistical analysis comparing the two arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.